CLINICAL TRIAL: NCT03163888
Title: Effects of Computer Navigation Versus Conventional Total Knee Arthroplasty on the Levels of Inflammation Markers: A Prospective Comparative Study
Brief Title: Effects of Navigation Versus Conventional Total Knee Arthroplasty on the Levels of Inflammation Markers
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 100-0038A3
Record Dates: First submitted 2017-05-11; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Arthroplasty Complications; Inflammatory Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling and collection of hemovac drainage after TKR surgeries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Navigation TKR group: TKR performed under computer navigation without violating distal femur bone marrow.
  Interventions: Procedure: Navigation TKR
- Conventional TKR group: TKR performed under conventional distal femur cutting juts with violation of distal femur bone marrow.

INTERVENTIONS:
Procedure: Navigation TKR — Traditional over Conventional TKR
  Groups: Navigation TKR group

SUMMARY:
Total knee arthroplasty (TKA) is a well-established modality for the treatment of advanced knee osteoarthritis with high satisfaction rate. However, the traditional cutting jigs for distal femur cutting inevitably violates the medullary canal of femoral bone. The process of intramedullary reaming for the insertion of distal femur cutting jigs stimulated the dissipation of marrow emboli that reported lead to increased risk of myocardial infarction or cardiac stress perioperatively. There are emerging refinements aiming to reduce the insult to the medullary canal of the distal femur as well as to improve the prosthetic alignment, such as navigation assisted TKA or robotic surgery.

In addition to better prosthetic alignment, computer-assisted navigation TKAs also mitigate perioperative blood loss and systemic emboli. The publication previously published by the investigators showed that navigation TKAs can lead to lesser extent of elevation of endothelial injury markers than the traditional TKAs. However, the detrimental effects of intramedullary reaming seem to be multi-dimensional and the whole picture has not been elucidated clearly at present.

Previous studies have shown that operative trauma can trigger marked immune responses. Operative procedures can simultaneously stimulate the pro-inflammatory and anti-inflammatory response, with 80% of the leucocyte transcriptome being affected. Most studies of hip or knee surgery found that operation-triggered immune reactions are associated with postoperative recovery, infection, and even mortality.

The navigation TKAs avoid the process of intra-medullary reaming, which is the mandatory part of conventional TKA for the distal femur cutting. The investigators hypothesize that the reaming process may exert substantial inflammatory response, which can be manifested by higher level of inflammatory markers in the serum and hemovac drainage samples obtained from the participants undergoing conventional TKAs.

ELIGIBILITY:
Inclusion Criteria:

* end stage knee OA necessitating TKR surgeries

Exclusion Criteria:

* autoimmune diseases, malignancies, previous knee surgery or post-traumatic arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients necessitating TKA surgery due to advanced degenerative osteoarthritis of the knee visited the outpatient department initially and were then scheduled for admission for TKA surgery. The patients were self-separated into two groups when they visited the outpatient department. The patients visiting professor CJ Wang would undergo conventional TKA, and those visiting Dr. JY Ko would undergo navigation TKA. Both senior authors had performed more than 1,000 TKAs using the conventional and navigation method respectively before recruiting the patients of our study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Concentration of IL-6(pg/mL) | 24 hours after TKR
  serum level change from baseline 24 hours after TKR , hemovac level 24 hours after TKR

SECONDARY OUTCOMES:
Concentration of IL-10(pg/mL) | 24 hours after TKR
  serum level change from baseline 24 hours after TKR , hemovac level 24 hours after TKR
Concentration of TNF-alpha (pg/mL) | 24 hours after TKR
  serum level change from baseline 24 hours after TKR , hemovac level 24 hours after TKR

IPD SHARING:
Plan to Share IPD: No